CLINICAL TRIAL: NCT02827305
Title: Clinical Evaluation of the Centella Asiatica (Gotukola) Mouthwash as an Adjunct to Mechanical Plaque Control: A RCT
Brief Title: Centella Asiatica (Gotukola) Mouthwash as an Adjunct to Mechanical Plaque Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sri Hasanamba Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Talat Mohammadi, Post graduate student, Sri Hasanamba Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDCH/2015-16/1409
Record Dates: First submitted 2016-05-13; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Gingival Diseases
Keywords: antiplaque; antigingivitis
MeSH Terms: conditions — Gingival Diseases | interventions — Centella asiatica extract; Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Experimental): scaling and Gotukola mouthwash intervention- 1.Scaling 2.Gotukola mouthwash , 10ml twice daily to be rinsed for 60 seconds
  Interventions: Drug: Gotukola; Procedure: Scaling
- group 2 (Active Comparator): Scaling
  Interventions: Procedure: Scaling
- group 3 (Active Comparator): Intervention- Gotukola mouthwash only is advised to be used two times a day, each time 10ml rinsed for 60 seconds (morning and evening ) after the food.
  Interventions: Drug: Gotukola

INTERVENTIONS:
Drug: Gotukola — 10 ml of mouthwash to be rinsed for duration of 60 seconds
  Other Names: Centella Asiatica
  Arms: group 1; group 3
Procedure: Scaling — Ultrasonic scaling was performed in one visit on both upper and lower arches.
  Arms: group 1; group 2

SUMMARY:
This study evaluates the adjunctive use of Centella Asiatica (gotukola) to scaling in the reduction of plaque and gingival inflammation. Patients were divided into three groups of which group 1 received scaling and gotukola mouthwash, group 2 received scaling only and group 3 received gotukola mouthwash only.

DETAILED DESCRIPTION:
Mechanical plaque control by tooth brushing is considered to be the ideal way of preventing plaque associated gingivitis. However due to various factors individuals fail to perform an adequate quality of self performed plaque control. Centella Asiatica (gotukola) possess wide range of biological activities like anti-inflammatory, anti-psoriatic, anti-ulcer, hepato-protective, anticonvulsant, immunostimulant, cardioprotective, antidiabetic, antiviral, antibacterial, antifungal, etc. So, it could be used as adjunctive to mechanical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 22 natural teeth
* Participants with Chronic generalized gingivitis
* Participants with plaque index score ≥1

Exclusion Criteria:

* Participants with fixed or removable appliances
* Participants with more than full coverage restorations
* Medically compromised participants
* Participants on long term medications
* Smokers
* Participants who had used any type of antibacterial mouthwash in 4weeks of commencement.
* Patients with history of recent periodontal therapy

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The efficacy of gotukola as an adjunct to scaling was assessed by using plaque index and gingival indes | 2-8-2015 to 16-8-2015
  A total of 36 patients were participated in the study and the outcome measures were assessed 15 days after the start of the study, PLaque index ( Silnes and Loe 1964) - The buccal, lingual,mesial and distal surfaces of the index teeth is given a scoring from 0-3 The scores from the four areas of the teeth are added and divided by four in order to give the plaque index of the tooth. The index for the patient is obtained by summing the indices for all six teeth and dividing by six. Gingival index -Loe and Silnes 1963- The buccal, lingual,mesial and distal surfaces of all ginival tissues of index teeth were given a scroe from 0-3.This then constitutes the GI for the area and scores from the 4 areas of the tooth are added and divided by four to give GI for the tooth. Scores for individual teeth may be grouped to designate the GI for the group of the teeth. The scores are added and divided by nu,ber of teeth to get GI for an individual

CONTACTS AND LOCATIONS:
Overall Officials: Talat Mohammadi, PG student, Principal Investigator — Sri Hasanamba Dental College and Hospital
Locations (1):
- Talat Mohammadi, Hassan, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sastravaha G, Yotnuengnit P, Booncong P, Sangtherapitikul P. Adjunctive periodontal treatment with Centella asiatica and Punica granatum extracts. A preliminary study. J Int Acad Periodontol. 2003 Oct;5(4):106-15. PMID 14604059
- [Background] Sastravaha G, Gassmann G, Sangtherapitikul P, Grimm WD. Adjunctive periodontal treatment with Centella asiatica and Punica granatum extracts in supportive periodontal therapy. J Int Acad Periodontol. 2005 Jul;7(3):70-9. PMID 16022023